CLINICAL TRIAL: NCT03212014
Title: Development and Research of an Individualized Intelligent Platform for Rehabilitaion in Patients With Parkinson's Disease
Brief Title: Development and Research of an Individualized Intelligent Platform for Rehabilitaion in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-09-018C
Record Dates: First submitted 2017-07-06; First posted 2017-07-11 (Actual); Last update posted 2017-07-11 (Actual); Status verified 2017-07

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; intelligent; Rehabilitaion
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LSVT-BIG (Experimental): Participants in this group would be treated with LSVT-BIG for three months
  Interventions: Other: LSVT-BIG
- POWER (Experimental): Participants in this group would be treated with POWER for three months
  Interventions: Other: POWER
- Traditional rehabilitation (Active Comparator): Participants in this group would be treated with traditional exercise rehabilitation for three months
  Interventions: Other: Traditional rehabilitation

INTERVENTIONS:
Other: LSVT-BIG — LSVT BIG can be delivered by a physical or occupational therapist. Treatment is administered in 16 sessions over a single month (four individual 60 minute sessions per week). This protocol was developed specifically to address the unique movement impairments for people with Parkinson disease. The protocol is both intensive and complex, with many repetitions of core movements that are used in daily living. This type of practice is necessary to optimize learning and carryover of your better movement into everyday life!
  Arms: LSVT-BIG
Other: POWER — Power Rehabilitation(PR), a new resistance training regime, can improve in power and independence level of the elderly people. The first word of PR was in brief of Produce Outcome Worthwhile for the Elderly Rehabilitation (POWER)
  Arms: POWER
Other: Traditional rehabilitation — traditional exercise models in currently clinical use
  Arms: Traditional rehabilitation

SUMMARY:
The present study aims to compare the clinical efficacy of intelligent POWER therapy, intelligent LSVT-BIG therapy, and the three exercise models currently in clinical use. DCM_IR analysis will also be incorporated into the analysis to develop a personalized and intelligent Parkinson's rehabilitative therapy platform.

DETAILED DESCRIPTION:
Background:

Parkinson's disease is a progressively degenerative disorder. Patients need early screening, therapeutic intervention, and personalized interaction with outpatient rehabilitative treatment. In the past, it had been difficult to meet these goals. Recent advances in bio-sensors technology has enabled collection of bio-metric data. Models of brainwave analysis have also matured. In addition, our ability to analyze vibrational spectrogram had also greatly improved. How to combine these enabling technologies to meet the needs of Parkinson's patients is an urgent topic of research.

Objective:

The present study aims to compare the clinical efficacy of intelligent POWER therapy, intelligent LSVT-BIG therapy, and the three exercise models currently in clinical use. DCM_IR analysis will also be incorporated into the analysis to develop a personalized and intelligent Parkinson's rehabilitative therapy platform.

Method:

Patients will be randomly assigned into three groups, i.e. intelligent POWER, intelligent LSVT-BIG, and current protocol group. Single blind data collection will be used. Patients will be evaluated immediately before treatment, immediately after treatment, and 4 weeks after treatment. Evaluated criteria will include mini-BESTest, Unified Parkinson's disease rating scale, muscle power of lower extremity, time up and go, walk velocity, step length, cadence, and Parkinson's disease questionnaire PDQ-39.

Expected Outcome:

An intelligent rehabilitative therapy platform may be built on the sensor data and neural-network analysis of the data. The platform will enable patients to interact with medical personnel on out-patient basis. If further combined with DCM_IR analysis, personalized therapeutic efficacy indicator may be uncovered, thereby, realizing intelligent personalized rehabilitative therapy.

ELIGIBILITY:
Inclusion Criteria:

1. .Parkinson's disease diagnosis, Hoehn-Yahr level I-III
2. .Stable medicine intake for 2 weeks at least
3. .Able to walk independently for 15 meters
4. .Aged 40-85 years old

Exclusion Criteria:

1. .Cognition deficits(MMSE score<24)
2. .Combined other neurological disease, such as stork, SCI, and so on.
3. .Pregnant or Breastfeeding

Ages: 40 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2017-12-31 (Estimated); Study Completion 2017-12-31 (Estimated)

PRIMARY OUTCOMES:
mini-BESTest | 15 mins
  Mini BESTest assesses dynamic balance, a unidimensinal construct and includes 14 items addressing 4 of the 6 sections of the original BESTest (anticipatory postural adjustments, reactive postural control, sensory orientation, dynamic gait).

SECONDARY OUTCOMES:
Unified Parkinson's disease rating scale | 15 mins
  The unified Parkinson's disease rating scale (UPDRS) is used to follow the longitudinal course of Parkinson's disease. The UPD rating scale is the most commonly used scale in the clinical study of Parkinson's disease.
muscle power of lower extremity | 5 mins
  Muscle power of knee flexion, extension. Measured by MicroFET
PDQ-39 | 30 mins
  The PDQ-39 is a 39-item self-report questionnaire, which assesses Parkinson's disease-specific health related quality over the last month

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospial, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2024 Apr 8;4(4):CD013856. doi: 10.1002/14651858.CD013856.pub3. PMID 38588457
- [Derived] Ernst M, Folkerts AK, Gollan R, Lieker E, Caro-Valenzuela J, Adams A, Cryns N, Monsef I, Dresen A, Roheger M, Eggers C, Skoetz N, Kalbe E. Physical exercise for people with Parkinson's disease: a systematic review and network meta-analysis. Cochrane Database Syst Rev. 2023 Jan 5;1(1):CD013856. doi: 10.1002/14651858.CD013856.pub2. PMID 36602886